CLINICAL TRIAL: NCT02830984
Title: Nasobiliary Drainage After Endoscopic Sphincterotomy Plus Large-balloon Dilation for Preventing Postoperative Pancreatitis in Treating of Large Bile Duct Stones
Brief Title: ENBD After Endoscopic Sphincterotomy Plus Large-balloon Dilation for Preventing PEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ENBD-001
Record Dates: First submitted 2016-07-09; First posted 2016-07-13 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2016-07

CONDITIONS: Post-ERCP Acute Pancreatitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EST+LBD+ENBD group (Experimental): Nasobiliary drainage after endoscopic sphincterotomy plus large-balloon dilation in treating of large bile duct stones
  Interventions: Procedure: EST+LBD+ENBD
- EST+LBD group (Active Comparator): Without nasobiliary drainage after endoscopic sphincterotomy plus large-balloon dilation in treating of large bile duct stones
  Interventions: Procedure: EST+LBD

INTERVENTIONS:
Procedure: EST+LBD+ENBD — Nasobiliary drainage after endoscopic sphincterotomy plus large-balloon dilation in treating of large bile duct stones
  Arms: EST+LBD+ENBD group
Procedure: EST+LBD — Without nasobiliary drainage after endoscopic sphincterotomy plus large-balloon dilation in treating of large bile duct stones
  Arms: EST+LBD group

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) has become one of the most important techniques in the treatment of bile duct stones. A number of studies have been conducted using large-balloon dilation (LBD) after adequate EST to extract large bile duct stones. In those studies, the authors suggested that EST plus LBD might lower the risk of post procedure pancreatitis (PEP) by directing balloon dilation toward the bile duct rather than the pancreatic duct. It has been reported that EPBD followed by insertion of nasobiliary drainage catheter can prevent PEP. However, it is still unclear that nasobiliary drainage after endoscopic sphincterotomy plus large-balloon dilation for preventing postoperative pancreatitis in treating of large bile duct stones.The investigators therefore designed a prospective randomized trial to determine whether nasobiliary drainage prevent PEP after endoscopic sphincterotomy plus LBD for the treatment of large bile duct stones.

DETAILED DESCRIPTION:
Patients enrolled were confirmed the presence of CBD stones using magnetic resonance cholangiopancreatography. Patients with large bile duct stones were randomly assigned to EST+LBD+ENBD group and EST+LBD group. A descriptive analysis will be performed on primary endpoint, containing frequency of number and percentage of patients. A two proportion equality test will be conducted to explore whether incidence rates are different. Descriptive statistics including number (N), mean, median, standard deviation, minimum and maximum, will be produced for all continuous variables. Frequency tables of number (N) and percentage of subjects will be produced for all categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients with visualized bile duct stones ≥12 mm in maximum transverse diameter. - Males and females, age > 18 years.
* Normal amylase level before undergoing ERCP.
* Signed inform consent form and agreed to follow-up on time.

Exclusion Criteria:

* Bleeding diathesis
* Prior EST or EPBD or ENBD
* Billroth II or Roux-en-Y anatomy
* Distal extrahepatic bile duct stenosis
* Acute pancreatitis
* Intrahepatic bile duct stones.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The prophylaxis effect of ENBD on post-ERCP pancreatitis after endoscopic sphincterotomy plus LBD for the treatment of large bile duct stones. | the incidence of post-ERCP pancreatitis at 24 h after ERCP in two groups
  If the serum amylase of patients elevation and 3 times higher than the normal values after ERCP 24 hours in high risk patients, who also have clinical symptoms, without other acute abdominal diseases,such as gastrointestinal perforation,acute cholecystitia and acute cholangitis and etc. In this condition, it will be defined PEP(post-ERCP pancreatitis).
  Descriptive statistics will be produced for all continuous variables. Frequency tables of number (N) and percentage of subjects will be produced for all categorical variables.

SECONDARY OUTCOMES:
Compare EST+LBD+ENBD group EST+LBD with group on the incidence of hyperamylasemia/adverse events. | the incidence of hyperamylasemia/adverse events at 24 h after ERCP in two groups
  Hyperamylasemia will be defined as the serum amylase 3 times more than the upper normal values, without clinical symptoms. During the study, any unexpected medical issue will be called adverse event.
  Descriptive statistics will be produced for all continuous variables. Frequency tables of number (N) and percentage of subjects will be produced for all categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Shao Feng, MD, Principal Investigator — Department of General Surgery, Anhui Provincial Hospital Affiliated with Anhui Medical University
Locations (1):
- Department of General Surgery, Anhui Provincial Hospital Affiliated with Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No